CLINICAL TRIAL: NCT01507467
Title: IAEA-HypoX. A Randomized Multicenter Study of Accelerated Fractionated Radiotherapy With or Without the Hypoxic Radiosensitizer Nimorazole in the Treatment of Squamous Cell Carcinoma of the Head and Neck
Brief Title: IAEA-HypoX. Accelerated Radiotherapy With or Without Nimorazole in Squamous Cell Carcinoma of the Head and Neck
Acronym: IAEA-HypoX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Danish Head and Neck Cancer Group (Network)
Collaborators: International Atomic Energy Agency (Other Government); Danish Center for Interventional Research in Radiation Oncology (CIRRO) (Other)
Responsible Party: Principal Investigator, Jens Overgaard, Professor, Danish Head and Neck Cancer Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAEA-HypoX; IAEA-HypoX (Other Grant/Funding Number: IAEA, CIRRO; Aarhus University, Denmark, AZANTA Denmark)
Record Dates: First submitted 2011-08-14; First posted 2012-01-11 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Head and Neck Carcinoma
Keywords: Head and neck carcinoma; Accelerated radiotherapy; Hypoxic modification with Nimorazole
MeSH Terms: interventions — Radiation; Nimorazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Accl. RT (Active Comparator): Accelerated Radiotherapy 66-70 Gy, 2Gy/fx, 6fx/week
  Interventions: Radiation: Accl. RT
- Accl. RT + Nimorazole (Experimental): Accelerated Radiotherapy 66-70 Gy, 2Gy/fx, 6fx/week + Nimorazole
  Interventions: Radiation: Accl. RT; Radiation: Accl. radiotherapy + Nimorazole

INTERVENTIONS:
Radiation: Accl. RT — Accelerated Radiotherapy: Radiotherapy 66-70 Gy, 2Gy/fx, 6fx/week
  Other Names: Radiation Oncology, Accelerated fractionation
Radiation: Accl. radiotherapy + Nimorazole — Radiation: Radiotherapy 66-70 Gy, 2Gy/fx, 6fx/week plus Nimorazole (tablets or powder) 1.2 g/m2 body surface in connection with the first daily radiation treatments
  Other Names: Hypoxic radiosensitizer, Nimorazole, Nimoral
  Arms: Accl. RT + Nimorazole

SUMMARY:
The purpose of this study is to test the hypothesis that radiotherapy of head and neck carcinoma can be improved by hypoxic modification of radiotherapy using nimorazole as a hypoxic radiosensitizer in association with accelerated fractionation, in an unselected patient population in a global environment.

DETAILED DESCRIPTION:
Squamous cell carcinoma in the head & neck region (HNSCC) accounts for approximately 7% of all cancers worldwide & around 75% of all HNSCC cases are seen in the less developed countries.

Significant improvement in loco-regional control & disease specific survival by radiation therapy could be achieved by reducing the overall treatment time by "Accelerated Fractionation" schedule.

Modification of hypoxia by Nimorazole demonstrated significant improved local effect of radiation with neither serious nor lasting side effects. So, it is expected that the optimal treatment option is reducing the overall treatment time with concomitant use of Nimorazole. Such treatment principle is optimal for testing in developing countries.

The aim of the study:

* To determine the possible therapeutic gain of using nimorazole given as a hypoxic radiosensitizer in conjunction with accelerated fractionated radiotherapy of invasive squamous cell carcinoma of the larynx, pharynx and oral cavity, and
* To determine whether the addition of Nimorazole to primary curative radiotherapy is feasible and tolerable on a worldwide scale.
* To evaluate the tolerance, compliance and toxicity of using nimorazole.

ELIGIBILITY:
Inclusion Criteria:

* Tumor classified as stage I-IV located in oropharynx, hypopharynx, larynx (not glottic stage I-II), or oral cavity according to the TNM classification.
* Histopathological diagnosis of invasive squamous cell carcinoma in the primary tumor.
* Informed consent according to the Helsinki declaration and local regula-tions.
* The patient must be candidate for external beam radical radiotherapy, and must be expected to accomplish the treatment.
* Performance status 0-2 according to WHO criteria.
* The patient should not have symptoms of peripheral neuropathy assessed by clinical examination.
* Normal function of liver and kidney by routine laboratory examinations. The patient must not be pregnant

Exclusion Criteria:

* Distant metastases.
* The patient should not be in a state or condition that could be expected to influence the outcome of treatment, or complicate the assessment or the treatment follow-up, or (apart from the present disease) reduce the life expectancy.
* Surgical excision (except biopsy), prior or planned (including elective neck dissection).
* The existence of synchronous multiple malignancies (not leukoplakia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Locoregional control after curative intended radiotherapy +/- Nimorazole | 5-years

SECONDARY OUTCOMES:
Disease specific survival | 5.years
Overall survival | 5-years
Treatment related morbidity | 5-years
  Treatment related acute and late morbidity releted to radiotherapy and/or nimorazole treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jens Overgaard, MD, Principal Investigator — Department of Experimental Clinical Oncology, Aarhus University Hospital, Denmark; Mohamed Hassan, MD, Study Director — Study Coordinator
Locations (6):
- Radiation Oncology Department, National Cancer Institute, Cairo, Egypt
- Radiation Oncology Center, Tallinn, Estonia
- Pakistan (3):
  - Nuclear Medicine, Oncology & Radiotherapy Institute, Radiation Oncology Department G-8/3, Islamabad
  - Karachi Institute of Radiotherapy and Nuclear Medicine, Karachi
  - Institute of Radiotherapy and Nuclear Medicine (IRNUM) Hospital Peshawar, Peshawar
- Institute of Oncology Department of Radiation Oncology, Ljubljana, Slovenia